CLINICAL TRIAL: NCT05398445
Title: A Phase 3, 24-week, Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy, Safety and Tolerability of Rocatinlimab (AMG 451) Monotherapy in Adult Subjects With Moderate-to-severe Atopic Dermatitis (AD)
Brief Title: A Study Evaluating Rocatinlimab in Moderate-to-severe Atopic Dermatitis (ROCKET-IGNITE)
Acronym: ROCKET-Ignite
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210142; 2022-501540-15-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AMG 451; KHK4083; Rocatinlimab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Rocatinlimab Dose 1 every 4 weeks (Q4W) + loading dose at Week 2
  Interventions: Drug: Rocatinlimab
- Arm B (Experimental): Rocatinlimab Dose 2 Q4W + loading dose at Week 2
  Interventions: Drug: Rocatinlimab
- Arm C (Placebo Comparator): Placebo Q4W+ loading dose at Week 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rocatinlimab — Participants will receive Rocatinlimab subcutaneously.
  Other Names: AMG 451
  Arms: Arm A; Arm B
Drug: Placebo — Participants will receive a placebo subcutaneously.
  Arms: Arm C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rocatinlimab in monotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with a diagnosis of AD according to the AAD Consensus Criteria (2014) present for at least 12 months
* History of inadequate response to TCS (Topical Corticosteroid) of medium to higher potency (with or without topical calcineurin inhibitors [TCI]).
* EASI score ≥16
* vIGA-AD score ≥3
* ≥10% body surface area (BSA) of AD involvement
* Worst pruritus numerical rating scale ≥ 4

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  * Systemic corticosteroids
  * Systemic immunosuppressants
  * Phototherapy
  * Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week, prior to Day 1:

  * TCS of any potency
  * TCI
  * Topical phosphodiesterase type 4 inhibitors
  * Other topical immunosuppressive agents
  * Combination topical agents including TCS of any potency, TCI, PDE4 inhibitors, or other topical immunosuppressive agents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Achievement of a Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) score of 0 or 1 with ≥2 point reduction from baseline at Week 24 | Baseline, Week 24
Achievement of ≥75% reduction from baseline in Eczema Area and Severity Index (EASI) score at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Achievement of ≥75% reduction from baseline in EASI score at Week 16 | Baseline, Week 16
Achievement of a vIGA-AD score of 0 or 1 from baseline at Week 16 | Baseline, Week 16
Achievement of a ≥ 4-point reduction from baseline in weekly average of daily worst pruritus numerical rating scale (NRS) score at Week 16 in subjects with baseline weekly average of daily worst pruritus NRS score ≥ 4 | Baseline, Week 16
Achievement of a ≥ 4-point reduction from baseline in weekly average of daily worst pruritus NRS score at Week 24 in subjects with baseline weekly average of daily worst pruritus NRS score ≥ 4 | Baseline, Week 24
Achievement of ≥90% reduction from baseline in EASI score at Week 24 | Baseline, Week 24
Achievement of a ≥ 4-point reduction from baseline in weekly average of daily AD skin pain NRS score at Week 24 in subjects with baseline weekly average of AD skin pain NRS score ≥ 4 | Baseline, Week 24
Achievement of a vIGA-AD 1 response with presence of only barely perceptible erythema or vIGA-AD 0 response (revised Investigator's Global Assessment [rIGA™] 0/1) at Week 24 | Baseline, Week 24
Achievement of Facial AD Severity Score (FASS) of clear at Week 24 for subjects with facial AD at baseline | Baseline, Week 24
Achievement of Hand AD Severity Score (HASS) of clear at Week 24 for subjects with hand AD at baseline | Baseline, Week 24
Change from baseline in weekly average of daily worst pruritus NRS score at week 16 | Baseline, Week 16
Change from baseline in weekly average of daily worst pruritus NRS score at Week 24 | Baseline, Week 24
Change from baseline in SCORing Atopic Dermatitis (SCORAD) itch visual analogue scale (VAS) score at Week 16 | Baseline, Week 16
Change from baseline in SCORAD itch VAS score at Week 24 | Baseline, Week 24
Achievement of ≥ 4-point reduction from baseline in DLQI score at Week 24 in subjects with baseline DLQI score ≥ 4 | Baseline, Week 24
Change from baseline in DLQI score at Week 24 | Baseline, Week 24
Achievement of ≥ 4-point reduction from baseline in POEM score at Week 24 in subjects with baseline POEM score ≥ 4 | Baseline, Week 24
Change from baseline in POEM score at Week 24 | Baseline, Week 24
Achievement of a ≥ 4-point reduction from baseline in weekly average of daily AD skin pain NRS score at Week 16 in subjects with baseline weekly average of AD skin pain NRS score ≥ 4 | Baseline, Week 16
Change from baseline in weekly average of daily AD skin pain NRS score at Week 24 | Baseline, Week 24
Change from baseline in weekly average of daily AD skin pain NRS score at Week 16 | Baseline, Week 16
Achievement of a ≥ 3-point reduction from baseline in weekly average of daily AD skin pain NRS score at Week 24 in subjects with baseline weekly average of AD skin pain NRS score ≥ 3 | Baseline, Week 24
Achievement of a ≥ 3-point reduction from baseline in weekly average of daily AD skin pain NRS score at Week 16 in subjects with baseline weekly average of AD skin pain NRS score ≥ 3 | Baseline, Week 16
Change from baseline in weekly average of daily sleep disturbance NRS score at Week 24 | Baseline, Week 24
Achievement of Hospital Anxiety and Depression Scale (HADS)-anxiety subscale score < 8 at Week 24 in subjects with baseline HADS-anxiety subscale score ≥ 8 | Baseline, Week 24
Change from baseline in HADS-anxiety subscale score at Week 24 | Baseline, Week 24
Achievement of HADS-depression subscale score < 8 at week 24 in subjects with baseline HADS-depression subscale score ≥ 8 | Baseline, Week 24
Change from baseline in HADS-depression subscale score at Week 24 | Baseline, Week 24
Achievement of a ≥ 8.7-point reduction from baseline in SCORAD score at Week 24 in participants with baseline SCORAD score ≥ 8.7 | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (202):
- United States (50):
  - Cahaba Dermatology and Skin Health Center, Birmingham, Alabama
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - First OC Dermatology, Fountain Valley, California
  - Kaiser Permanente - Glendale Medical Center, Glendale, California
  - Long Beach Research Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Cura Clinical Research, Sherman Oaks, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Skin Care Research Incorporated, Boca Raton, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - Global Research Associates, Homestead, Florida
  - Healthy Life Research, Miami, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Kirsch Dermatology LLC, Naples, Florida
  - Pure Skin Dermatology and Aesthetics, Orlando, Florida
  - Industrial Medicine Associates Ima Clinical Research Inc, St. Petersburg, Florida
  - Genesis Clinical Research LLC, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - DeNova Research, Chicago, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - The Indiana Clinical Trials Center PC, Plainfield, Indiana
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Onyx Clinical Research, Flint, Michigan
  - Dermatology and Skin Cancer Center of Lees Summit, Lee's Summit, Missouri
  - Jubilee Clinical Research Inc, Las Vegas, Nevada
  - Allcutis Research, Llc - Portsmouth, Portsmouth, New Hampshire
  - Continental Clinical Solutions - Cherry Hill, Cherry Hill, New Jersey
  - Industrial Medicine Associates Ima Clinical Research Inc, Hartsdale, New York
  - Sadick Research Group, New York, New York
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - The Skin Surgery Center for Clinical Research, Winston-Salem, North Carolina
  - Optima Research, Boardman, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Dermatology Research Center of Oklahoma, PLLC, Tulsa, Oklahoma
  - Essential Medical Research LLC, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - DermDox Dermatology, LLC, Sugarloaf, Pennsylvania
  - Cumberland Skin Center, Hermitage, Tennessee
  - Dermatology Treatment and Research Center PA, Dallas, Texas
  - The Woodlands Dermatology Associates, The Woodlands, Texas
  - Education and Research Foundation Inc, Lynchburg, Virginia
  - Frontier Derm Partners, Mill Creek, Washington
  - West Virginia Research Institute, Morgantown, West Virginia
- Argentina (9):
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Fundacion Respirar, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Derqui, Pilar, Buenos Aires
  - Centro Dermatológico Schejtman, San Miguel, Buenos Aires
  - InAER - Investigaciones en Alergia y Enfermedades Respiratorias, Buenos Aires, Distrito Federal
  - Instituto de Neumonologia y Dermatologia, Buenos Aires, Distrito Federal
  - Conexa Investigacion Clinica SA, CABA, Distrito Federal
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Diagnostico Abc American British Cowdray, Rosario, Santa Fe Province
- Brazil (8):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Upeclin-Pesq Clin FacMed Botucatu, Botucatu, São Paulo
  - Hosp e Maternidade Dr Christovao da Gama, Santo André, São Paulo
  - Fundacao Abc - Centro Univ Fmabc, Santo André, São Paulo
  - Consultoria Medica e Pesquisa Clinica Cmpc, Sorocaba, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Alergoalfa Nucleo Diagnostico Tratamento e Pesquisa Clinica em Alergia, São Paulo
- Canada (12):
  - Alberta Derma Surgery Centre, Edmonton, Alberta
  - Vida Clinical Research, Edmonton, Alberta
  - CCA Medical Research Corporation, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - LEADER Research, Hamilton, Ontario
  - DermEdge Research Incorporated, Mississauga, Ontario
  - Canadian Dermatology Centre, North York, Ontario
  - Gordon Sussman Clinical Research Incorporated, North York, Ontario
  - Oak Ridges Aesthetics Centre, Richmond Hill, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Recherche Clinique Sigma Incorporated, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- China (23):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital ,Sun-Yat Sen University, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First Peoples Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Union Hospital Tongji Medical College Huazhong University of science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangyin Hospital of Traditional Chinese Medicine, Jiangyin, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - the First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Affiliated Hangzhou First Peoples Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Peking University Peoples Hospital, Beijing
  - Shanghai Skin Disease Hospital, Shanghai
- Croatia (3):
  - Special Hospital for Medical Rehabilitation Naftalan, Ivanić-Grad
  - Sestre milosrdnice University Hospital Center, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (7):
  - Dermamedica, sro, Náchod
  - CCR Ostrava sro, Ostrava
  - Pratia Pardubice as, Pardubice
  - Clintrial sro, Prague
  - Pratia Prague sro, Prague
  - Fakultni nemocnice Bulovka, Prague
  - Krajska zdravotni as - Masarykova nemocnice Usti nad Labem oz, Ústí nad Labem
- Germany (12):
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Dermatologische Gemeinschaftspraxis-Mahlow, Blankenfelde-Mahlow
  - Hautarztpraxis Dr Niesmann und Dr Othlinghaus, Bochum
  - Rosenpark Research GmbH, Darmstadt
  - Universitaetsklinikum Dresden, Dresden
  - Heinrich-Heine-Universitaet Duesseldorf - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Essen, Essen
  - Institute for Health Services Research in Dermatology and Nursing, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Hautarztpraxis Dres Leitz und Kollegen, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
  - CentroDerm GmbH, Wuppertal
- Greece (7):
  - Athens Naval Hospital, Athens
  - Thoracic General Hospital Of Athens Sotiria, Athens
  - University General Hospital Attikon, Athens
  - Andreas Syngros Hospital Of Venereal And Dermatological Diseases, Athens
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - Papageorgiou General Hospital, Thessaloniki
- Medmare Bt, Veszprém, Hungary
- Italy (5):
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (19):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Central Clinic, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Matsuo Clinic, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Kaji Dermatology Clinic, Nonoichi-shi, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Takeoka Dermatology Clinic, Marugame-shi, Kagawa-ken
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Mochida Dermatology Clinic, Izumiotsu-shi, Osaka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
- Latvia (3):
  - Outpatient clinic Veselibas Centrs 4, Riga
  - Outpatient clinic Veselibascentrs 4, Riga
  - Smite Aija practice in dermatology and venerology, Talsi
- PreCare Trial and Recruitment, Born, Netherlands
- Poland (10):
  - AKK Medical Spolka z ograniczona odpowiedzialnoscia Centrum Medyczne Tu sie leczy, Gdansk
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Zdrowia i Urody Maxxmed, Lublin
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Spzoo, Malbork
  - Twoja przychodnia Ncm, Nowa Sól
  - Twoja przychodnia Pcm, Poznan
  - Twoja Przychodnia Scm, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Spzoo, Tarnów
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Dermatologiczna Praktyka Lekarska Michal Torz Dermaceum Centrum Badan Klinicznych, Wroclaw
- Portugal (4):
  - Hospital Lusiadas Lisboa, Lisbon
  - Hospital Cuf Descobertas, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
- Clinical Research of Puerto Rico, San Juan, Puerto Rico
- Slovakia (5):
  - Fakultna Nemocnica s poliklinikou F D Roosevelta Banska Bystrica, Banská Bystrica
  - Derma therapy, spol s ro, Bratislava
  - Sanare spol sro, Svidník
  - Kaderma Majtan, sro, Topoľčany
  - Fakultna nemocnica Trnava, Trnava
- South Korea (6):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - The Catholic University of Korea Incheon St Marys Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - National Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Clinico Universitario de Santiago, Pontevedra, Galicia
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- [Derived] Guttman-Yassky E, Kabashima K, Worm M, Luna PC, Hong HC, Chovatiya R, Bernstein JA, Kern JS, Ehst BD, Magnolo N, Herranz-Pinto P, Stein Gold L, Sofen H, Pink AE, Esfandiari E, Arai T, Yang Y, Shi R, Barragan C, Kricorian G, Schwartz-Sagi L, Bissonnette R. Efficacy and safety of rocatinlimab for the treatment of moderate-to-severe atopic dermatitis in ROCKET-IGNITE and ROCKET-HORIZON: two global, double-blind, placebo-controlled, randomised phase 3 clinical trials. Lancet. 2026 Jan 3;407(10523):53-66. doi: 10.1016/S0140-6736(25)01865-3. Epub 2025 Nov 25. PMID 41314226
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com